CLINICAL TRIAL: NCT01997177
Title: Assessment of Competence in Colonoscopy Using Motion Capture
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Preisler, MD, Rigshospitalet, Denmark
Other Study IDs: motion capture in colonoscopy
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Sensitivity Training Groups
Keywords: simulation; training; colonoscopy; standard setting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- novices: novice endoscopists, fellows of gastroenterology
- experienced endoscopist: consultant doctors of gastroenterology

SUMMARY:
Aim: To study the basic technical skills of colonoscopy using a MS Kinect for motion analysis. In order to develop a non-biased tool to monitor competence.

DETAILED DESCRIPTION:
To compare a group of novices to a group of experienced endoscopists performining colonoscopy.

Analyzing the motion pattern of the performers using a Kinect. Use the contrasting group method to set standards.

ELIGIBILITY:
Inclusion Criteria: none experience in colonoscopy or experience more than 350 colonoscopy procedures -

Exclusion Criteria: none

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctors in gastroenterology
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
to identify metrics of importans in colonoscopy training program | 3 months
  testing colonoscopy competence in a simulation lab. Finding metrics with discriminatory ability.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Preisler, MD, Principal Investigator — CEKU, Centre of clinical education, University of Copenhagen
Locations (1):
- CEKU, Centre of Clinical education, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Preisler L, Sondergaard Svendsen MB, Sondergaard B, Brink L, Nordentoft T, Svendsen LB, Konge L. Automatic and unbiased assessment of competence in colonoscopy: exploring validity of the Colonoscopy Progression Score (CoPS). Endosc Int Open. 2016 Dec;4(12):E1238-E1243. doi: 10.1055/s-0042-118226. Epub 2016 Nov 17. PMID 27995182